CLINICAL TRIAL: NCT02945332
Title: Incentivizing Lifestyle Modification to Reduce Disease Burden.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: RGK Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109495
Record Dates: First submitted 2016-08-31; First posted 2016-10-26 (Estimated); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Diabetes Mellitus
Keywords: exercise; activity; behavior
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Motor Activity; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Required supervised walking (Experimental): Device: Fitbit Flexes
  Interventions: Behavioral: Required supervised walking; Device: Fitbit Flex
- Non-required supervised walking (Active Comparator): Device: Fitbit Flexes
  Interventions: Behavioral: Non-required supervised walking; Device: Fitbit Flex

INTERVENTIONS:
Behavioral: Required supervised walking — The intervention will include meeting at an agreed upon community center location and time convenient for both the participant and the researcher. During these meetings, the participants will engage in indoor walking under the supervision of the researcher. This is to ensure accurate walking distance recording and also to monitor the participants for any potential adverse events. The participants will have the option of walking as long or short as they please, so long that it is less than 20 miles per week. This is to protect the participants from exhaustion or overexertion. Overall activity of this group will be recorded using Fitbit Flexes, worn at all time for the duration of the study.
  Arms: Required supervised walking
Behavioral: Non-required supervised walking — The intervention will include meeting at an agreed upon community center location and time convenient for both the participant and the researcher. During these meetings, the participants will engage in indoor walking not necessarily under the supervision of the researcher. Accurate walking distance recording will be done and also monitor the participants for any potential adverse events. The participants will have the option of walking as long or short as they please, so long that it is less than 20 miles per week. This is to protect the participants from exhaustion or overexertion. Overall activity of this group will be recorded using Fitbit Flexes, worn at all time for the duration of the study.
  Arms: Non-required supervised walking
Device: Fitbit Flex

SUMMARY:
Specifically, the main objective of this pilot and feasibility study is to develop the infrastructure that will be used in a larger study that would be proposed at a later date. Hence, this study has two parts. Part A: To establish contacts, collaboration, and networking to develop the infrastructure needed to conduct the study, Part B: To recruit eight subjects (4 subjects randomly assigned to either a control group or intervention group) from a low-income community in East Lubbock who are willing and able to participate in this pilot study. The research team's central hypothesis is that the disease burden of obesity and related co-morbidities could be attenuated within low-income communities by providing incentive-based free access to a safe and convenient exercise facility and earned credit to subsidize healthful food cost. The research team's secondary hypothesis is that the anticipated decrease in disease burden will make the incentivized changes in lifestyle cost-effective.

DETAILED DESCRIPTION:
Intervention Group:

After successfully passing the screening criteria, name, address, contact information, body weight (in light outdoor clothes and without shoes), height (without shoes), body fat percentage, BMI, waist circumference, age, and sex will be noted. Only the questions about medical history that are pertinent to determining the eligibility (as described above), will be asked. There will be a two week lead-in time period during which grocery store receipts will be collected and the participants will wear a Fitbit Flex pedometer at all times. This is to track food purchasing and consumption patterns and a method of determining a baseline activity level, respectively. The participants will meet with the researcher at the beginning of this two week period in order to give the participants the Fitbit Flexes. These receipts will be collected at the end of the two week time period.

After this lead-in, the participants will begin their four week testing period. Body weight and body fat will be determined on day 0 by using a bioimpedance measurement scale. This is a scale like the bathroom scale on which a person stands and holds onto two handles connected to the base by cables, while the machine reads body weight and body fat content (by passing a mild electric current through the body, similar to an electrocardiogram). Body weight and fat content will be determined once per week, for 4 weeks. The last body weight and body fat measurements will be at the end of the 4 week walking period. The four week testing period will include meeting at an agreed upon community center location and time convenient for both the participant and the researcher. During these meetings, the participants will engage in indoor walking under the supervision of the researcher. This is to ensure accurate walking distance recording and also to monitor the participants for any potential adverse events. The participants will have the option of walking as long or short as they please, so long that it is less than 20 miles per week. This is to protect the participants from exhaustion or overexertion. This process will continue for four weeks. At the end of each week, grocery store receipts will be collected to reflect food purchasing and consumption. The Fitbit Flex will remain worn by the participants at all times in order to track activity changes, outside of the supervised walking. At the end of this four week testing period, the total number of miles will be calculated (maximum of 80 miles). For every mile walked, the participants will earn dollar points. The money earned by each participant will be split between their utility payments and healthy food at a local grocery store. The research team will provide a list of healthful foods to the participants. It will include healthful foods such as fruits (and 100% juices), vegetables (and 100% juices), non-fat or low fat dairy products, low-fat whole grain products (bread, bagels, breakfast cereals, muffins), and uncooked fish and chicken.

During week 1, nutrition information will be provided. This will consist of brief nutrition information sessions and a grocery store tour to assist with selection of foods available with program coupons. The tour will be aimed at helping the subjects identify healthier food choices and to suggest alternatives and options to high-fat and/or low nutrient-dense foods.

After this four week testing period, there will be a secondary four week follow-up period. This will be the same as the four week testing period, minus the supervised walking and earning of money based on miles walked. This follow-up period is purposed to record food purchasing and consumption patterns along with everyday activity after their intervention. The participants will remain wearing their Fitbit Flexes and turning in their grocery store receipts.

Control Group:

The control group will have the same two week lead-in period in order to get a baseline food and activity level.

During the four week testing period for the control group, the participants will be encouraged to participate in supervised walking. However, the participants will not be earning money based on miles walked. The number of miles will be recorded, but strictly to be compared against the testing period of the intervention group.

The four week follow-up time period will be the same as the intervention group, with one exception. The control group will have the option to walk under supervision during their follow-up period in order to earn money under the same set of rules as the intervention group during their testing period. This opportunity to earn money is an effort to encourage participation and keep participants in the control group interested. The participants of the control group during the follow-up period will; however, continue to wear their Fitbit Flexes at all times and grocery store receipts will be collected.

Additional Procedural Information Throughout the study for both groups, the participants will be paid a small amount for their participation in the study. The payment will be identical for both the control and intervention groups. This is just a payment for the participants' time invested in the study. However, the participants will not receive their weekly participation money unless they turn in their receipts. This is to encourage the turning in of receipts for our study records.

In the prior arrangement with designated grocery stores, foods that could be purchased with the coupons or gift cards will be predetermined. The value, types of food, quantity purchased, and the user name will be recorded for further analysis.

At the end of the four week follow-up period for both groups, there will be an exit interview for all participants of the study. This interview will ask simple questions such as what the participants liked the most about the study, what they liked least, what we could improve upon, how they prefer to receive their earned money, and what most motivated them to walk. This interview will be one-on-one with the researcher and results will be kept confidential.

Text message reminders will be given in order to remind the participants of any upcoming appointments related to the study.

At the conclusion of the study for both groups, the participants will turn in their Fitbit Flexes to the researcher. The conclusion of this study for both groups will be the ten week mark, starting with the first day of the lead-in period and concluded at the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Sedentary (< 3 hours/week of moderate intensity physical activity), and otherwise healthy men and women
2. Willingness to: follow the instructions, and to attend regularly,
3. BMI 25 - 50 kg/M2
4. Age: 18y - 65 y. Subjects will be screened prior to the study.

Exclusion Criteria:

1. Significant cardiac disease in the past 6 months (Myocardial Infarction, angioplasty, Congestive Heart Failure, Left Bundle Branch Block, 3rd degree AV- block, CABG),
2. Uncontrolled hypertension (systolic BP > 180 or diastolic BP > 105 mm Hg),
3. Medications that could interfere with outcomes and that could not be safely withdrawn prior to testing,
4. Pregnancy or intention to conceive during the study period,
5. Current substance abuse,
6. Indications of potential difficulties adhering to the protocol,
7. Subjects who in the opinion of the investigators are inappropriate for study participation or who would be at additional risk by participating,
8. Physical or medical limitation for exercise, intermittent claudication, severe back pain or spasm, inability to ambulate independently or without the use of a cane or walker,
9. Unexcused absence for more than 2 continuous weeks, irregular attendance, non-cooperation, conception, or change in the health status that would jeopardize the subject could be grounds for expulsion from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lubbock Dream Center, Lubbock, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done by word of mouth and flyer, as only 8 subjects were required. Researchers connected with community/church leaders in the neighborhood to plan the recruitment of subjects for the study.
Pre-assignment Details: In total, 13 people were assessed. Four did not meet inclusion criteria, and 1 declined. Eight were enrolled. Subjects were given anonymous identifiers, subject IDs numbered 1-8. Randomization was completed as one-big-block-of-8. Four were chosen to be in the control group; the others received the intervention.
Groups:
- Required Supervised Walking: Device: Fitbit Flexes
  Required supervised walking: The intervention will include meeting at an agreed upon community center location and time convenient for both the participant and the researcher. During these meetings, the participants will engage in indoor walking under the supervision of the researcher. This is to ensure accurate walking distance recording and also to monitor the participants for any potential adverse events. The participants will have the option of walking as long or short as they please, so long that it is less than 20 miles per week. This is to protect the participants from exhaustion or overexertion. Overall activity of this group will be recorded using Fitbit Flexes, worn at all time for the duration of the study.
  Fitbit Flex
- Non-required Supervised Walking: Device: Fitbit Flexes
  Non-required supervised walking: The intervention will include meeting at an agreed upon community center location and time convenient for both the participant and the researcher. During these meetings, the participants will engage in indoor walking under the supervision of the researcher. This is to ensure accurate walking distance recording and also to monitor the participants for any potential adverse events. The participants will have the option of walking as long or short as they please, so long that it is less than 20 miles per week. This is to protect the participants from exhaustion or overexertion. Overall activity of this group will be recorded using Fitbit Flexes, worn at all time for the duration of the study.
  Fitbit Flex
Period: Overall Study
Arm/Group | Required Supervised Walking | Non-required Supervised Walking
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Required Supervised Walking | Non-required Supervised Walking | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Miles Walked
Description: This study will determine the miles walked in presence and absence of financial incentive
Time Frame: Conclusion of data recording; approximately 10 weeks after the participant begins the study.
Measure: Mean (Standard Error); unit: Miles
Groups:
- Non-required Supervised Walking: Device: Fitbit Flexes
  Non-required supervised walking: The intervention will include meeting at an agreed upon community center location and time convenient for both the participant and the researcher. During these meetings, the participants will engage in indoor walking not necessarily under the supervision of the researcher. Accurate walking distance recording will be done and also monitor the participants for any potential adverse events. The participants will have the option of walking as long or short as they please, so long that it is less than 20 miles per week. This is to protect the participants from exhaustion or overexertion. Overall activity of this group will be recorded using Fitbit Flexes, worn at all time for the duration of the study.
  Fitbit Flex
Arm/Group | Required Supervised Walking | Non-required Supervised Walking
Number analyzed (Participants) | 4 | 4
Miles | 1.1 (0.4) | 6.06 (3.6)
Statistical Analysis 1: Comparison: Required Supervised Walking vs Non-required Supervised Walking; Test type: Superiority; p = 0.32, Mixed Models Analysis; Mean Difference (Net) = 4.35, Standard Error of Mean 4.85

2. Secondary Outcome: Weight Change
Description: Weight will be recorded on an Omron portable bioimpedance scale.
Time Frame: From day 0 through week 6 of the study.
Measure: Mean (Standard Deviation); unit: Pounds (lbs)
Arm/Group | Required Supervised Walking | Non-required Supervised Walking
Number analyzed (Participants) | 4 | 4
Pounds (lbs) | 2.6 (3.0) | 0.8 (1.6)
Statistical Analysis 1: Comparison: Required Supervised Walking vs Non-required Supervised Walking; Test type: Superiority; p = 0.93, Mixed Models Analysis

3. Secondary Outcome: Body Fat Percentage Change
Description: Body fat percentage will be recorded with the Omron portable bioimpedance scale.
Time Frame: From day 0 through week 6 of the study.
Measure: Mean (Standard Deviation); unit: Change in percentage of body fat
Arm/Group | Required Supervised Walking | Non-required Supervised Walking
Number analyzed (Participants) | 4 | 4
Change in percentage of body fat | 1.3 (3.1) | 3.5 (6.9)
Statistical Analysis 1: Comparison: Required Supervised Walking vs Non-required Supervised Walking; Test type: Superiority; p = 0.16, Mixed Models Analysis; Mean Difference (Net) = 4.79, Standard Error of Mean 3.68

4. Secondary Outcome: Fat Mass Change
Description: Fat mass change will be recorded by the portable Omron bioimpedance scale.
Time Frame: From day 0 through week 6 of the study.
Measure: Mean (Standard Deviation); unit: Pounds (lbs)
Arm/Group | Required Supervised Walking | Non-required Supervised Walking
Number analyzed (Participants) | 4 | 4
Pounds (lbs) | 4.8 (6.9) | 0.15 (0.8)
Statistical Analysis 1: Comparison: Required Supervised Walking vs Non-required Supervised Walking; Test type: Superiority; p = 0.40, Mixed Models Analysis; Mean Difference (Net) = 11.36, Standard Error of Mean 15.32

5. Secondary Outcome: Fat Free Mass Change
Description: Fat free mass will be recorded with the Omron portable bio-impedance scale.
Time Frame: From day 0 through week 6 of the study.
Measure: Mean (Standard Deviation); unit: Pounds (lbs)
Arm/Group | Required Supervised Walking | Non-required Supervised Walking
Number analyzed (Participants) | 4 | 4
Pounds (lbs) | -2.15 (5.1) | 2.8 (3.9)
Statistical Analysis 1: Comparison: Required Supervised Walking vs Non-required Supervised Walking; Test type: Superiority; p = 0.77, Mixed Models Analysis; Mean Difference (Net) = -8.03, Standard Error of Mean 31.36

6. Secondary Outcome: Waist Circumference Change
Description: Waist circumference will be recorded with a body circumference tape.
Time Frame: From day 0 through week 6 of the study.
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | Required Supervised Walking | Non-required Supervised Walking
Number analyzed (Participants) | 4 | 4
Inches | 0.8 (2.0) | 0.7 (2.1)
Statistical Analysis 1: Comparison: Required Supervised Walking vs Non-required Supervised Walking; Test type: Superiority; p = 0.42, Mixed Models Analysis; Mean Difference (Net) = 2.98, Standard Error of Mean 4.16

7. Other Pre Specified Outcome: Food Purchasing Change
Description: This was a pre-specified outcome measure, but was not collected due to lack of availability of this data as this study did not collect food purchase receipts.
Time Frame: Day 0-6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were assessed every one month. There was no reported adverse event in the study.
Description: This study did not involve high risk. Walking was supervised and took place in a local community center. Participants had the option to immediately stop walking if they felt uneasy during walking. If it became apparent that the extent of an adverse event was beyond the research team's ability to handle, 911 would have been dialed immediately. The IRB would have been notified if any adverse event occurred.
Arm/Group | Required Supervised Walking | Non-required Supervised Walking
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No